CLINICAL TRIAL: NCT06760572
Title: Airway Data Collection With the Entarik Feeding Tube System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CRD-04-1877-01; R44AG076248 (NIH)
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Feeding Tube; feeding tube placement safety; feeding tube placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Healthy Adults (Experimental): Airway insertion
  Interventions: Device: Airway insertion

INTERVENTIONS:
Device: Airway insertion — Tube will be inserted into the trachea to make airway data measurements.

SUMMARY:
The purpose of this study is to evaluate the airway detection performance of the Entarik Feeding Tube System, and to collect data when the Entarik Feeding Tube is in the Airway for device development.

DETAILED DESCRIPTION:
The study is a prospective, single center, non-blinded, single arm study. Subjects who are scheduled to undergo an elective bronchoscopy procedure will have an Entarik Feeding Tube placed into the airway through an endotracheal tube under direct visualization while temperature and impedance data are collected by the Entarik monitor. Other data will be passively simultaneously collected through the Feeding Tube.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Able to provide informed consent.
3. Adults scheduled to undergo a bronchoscopy procedure who will be intubated as part of the standard of care.

Exclusion Criteria:

1. Known major upper airway malformation.
2. Presence of clinically significant respiratory infection.
3. Known bleeding disorder.
4. Currently pregnant.
5. Current basilar skull fracture.
6. Known sensitivities or allergies to the feeding tube components.
7. Deemed unsuitable for enrollment in study by the investigator based on subject's history (e.g., active anticoagulation therapy) or physical examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of accurate airway verifications by the Entarik feeding tube system | During the airway placement procedure
  Percentage of accurate verifications of airway placement of the tip of the Entarik feeding tube at the Safety Check Depth.
Incidence of Adverse Events | During the airway placement procedure
  Incidence of adverse events: (a) related to placement and (b) throughout the duration of the presence of the feeding tube within the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Burnett, MD, Study Director — Theranova, LLC
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographics and Primary Endpoint results.